CLINICAL TRIAL: NCT06704555
Title: A Study of the Radiotherapy Followed by Tiselizumab Combined With RCHOP in the Frontline Treatment of Follicular Lymphoma Patients With Bulky Disease
Brief Title: Radiotherapy Followed by Tiselizumab Combined With RCHOP in Previously Untreated Bulky Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-IIT02
Record Dates: First submitted 2024-11-12; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Follicular Lymphoma
Keywords: FL; Tiselizumab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Radiotherapy; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Treatment arm (Experimental): Radiation (dose:18～24Gy) ，chemoimmunotherapy 1～2 weeks later than radiation. Tiselizumab (200 mg iv d1) R-CHOP (rituximab 375 mg/m2 intravenous [IV] day 2, cyclophosphamide 750 mg/m2 IV day 3, doxorubicin 50 mg/m2 IV day 3, vincristine 1.4 mg/m2 [maximum 2.0 mg total] IV day 3, and prednisone 100 mg oral days 3-7, 21～28 days for one cycle ) for six cycles.
  Rituximab was given every 2 months to patients who were complete metabolic response /partial metabolic response（CMR/PMR）after first-line chemo until 2 years.
  Interventions: Radiation: radiation therapy; Drug: Tiselizumab; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Radiation: radiation therapy — received radiation (dose:18～24Gy)
Drug: Tiselizumab — 200 mg iv day 1
Drug: Rituximab — 375 mg/m2 intravenous [IV] day 2
Drug: Cyclophosphamide — 750 mg/m2 IV day 3
Drug: Doxorubicin — 50 mg/m2 IV day 3
Drug: Vincristine — 1.4 mg/m2 [maximum 2.0 mg total] IV day 3
Drug: Prednisone — 100 mg oral days 3-7

SUMMARY:
This was a single center, single arm, phase II study. Patients with previously untreated follicular lymphoma were enrolled from the department of lymphoma, Tianjin Medical University Cancer Institute and Hospital. The bulky disease was received radiation (dose:18～24Gy) before RCHOP. Patients began chemoimmunotherapy 1～2 weeks later than radiation. Treatment included Tiselizumab (200 mg iv d1) plus R-CHOP (rituximab 375 mg/m2 intravenous [IV] day 2, cyclophosphamide 750 mg/m2 IV day 3, doxorubicin 50 mg/m2 IV day 3, vincristine 1.4 mg/m2 [maximum 2.0 mg total] IV day 3, and prednisone 100 mg oral days 3-7, 21～28 days for one cycle ) for six cycles. Rituximab was given every 2 months to patients who were complete metabolic response /partial metabolic response（CMR/PMR）after first-line chemo until 2 years. Response was assessed by PET/CT scan after cycle 4 and cycle 6.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 positive (+) follicular lymphoma, grade 1, 2, or 3a，bulky disease (Mass diameter ≥ 7 cm)
* Have had no prior systemic treatment for lymphoma
* Meeting Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria for initiation of treatment
* Age 18-75 years
* ECOG Performance Status of 0-2 .Stage II, III, or IV by Ann Arbor staging system.
* Demonstrate adequate organ function as defined below; all screening labs to be obtained within 28 days prior to registration.

  1. Hematological: WBC≥3.5×109/L, Platelets ≥ 75×109/L,Absolute Neutrophil Count (ANC) ≥ 1.0×109/L，Hemoglobin (Hgb) ≥ 80 g/L
  2. Renal: Calculated creatinine clearance ≥ 50 mL/min
  3. Hepatic: Bilirubin ≤ 1.5 × upper limit of normal (ULN), AST/ALT ≤ 2.5×ULN
* Females of childbearing potential must be willing to abstain from vaginal intercourse or use an effective method(s) of contraception from the time of informed consent, during the study and for 6 months after the last dose of study drug(s). Males able to father a child must be willing to abstain
* Life expectancy ≥6 months
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Known active central nervous system lymphoma or leptomeningeal disease,
* Evidence of diffuse large B-cell transformation
* Grade 3b FL
* Concurrent malignancy or malignancy within the last 3 years (except for ductal breast cancer in situ, non-melanoma skin cancer, prostate cancer not requiring treatment, and cervical carcinoma in situ) whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial
* Known history of human immunodeficiency virus (HIV), or active hepatitis C Virus, or active hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed John Cunningham (JC) virus infection，any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association functional classification. Or left ventricular ejection fraction <50%;
* Known history of human immunodeficiency virus (HIV), or active hepatitis C Virus, or active hepatitis B Virus infection, or any uncontrolled active significant infection
* Known pneumonia associated with idiopathic pulmonary fibrosis, machine (for example, occlusive bronchiolitis), history of drug induced pneumonia, or screening during the chest computed tomography (CT) showed active pneumonia
* Have serious neurological or psychiatric history, can't normal study, including dementia, epilepsy, severe depression and mania
* Patients who were deemed by the investigator to be ineligible for enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Best Complete response (CR) rate | Through completion of treatment (estimated to be 2.5 year)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Best overall response rate (ORR) | Through completion of treatment (estimated to be 2.5 year)
  Objective Response rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
2 year progression-free survival | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The date of enrollment until disease progression or death from any cause.
Percentage of Participants With Adverse Events | Up to 30 days after completion of study treatment
  Adverse Events will be determined and graded on the basis of investigator assessments according to NCI CTC AE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided